CLINICAL TRIAL: NCT00309764
Title: Improving CHF Outcomes Through Interactive Voice Recognition (IVR) Data Acquisition and Targeted Nurse Follow-Up
Brief Title: CHF Management Using Telemedicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Project # 041873
Record Dates: First submitted 2006-03-31; First posted 2006-04-03 (Estimated); Last update posted 2006-04-03 (Estimated); Status verified 2006-03

CONDITIONS: Congestive Heart Failure (CHF)
MeSH Terms: conditions — Heart Failure | interventions — Telemedicine

INTERVENTIONS:
Behavioral: Telemedicine

SUMMARY:
The overall objective of this study is to improve clinical outcomes and quality of life for congestive heart failure (CHF) patients by integrating a readily available, low cost technology - the telephone - into coordinated CHF care.

DETAILED DESCRIPTION:
Strong patient-provider communication and vigilant home-based monitoring can be critical elements of successful chronic disease management. Among CHF patients, automated clinical data acquisition via the telephone can improve insight into inappropriate use of medications and onset of fluid overload or edema - indicating deteriorating heart function (notably worsening ejection fraction). Routine, timely monitoring of this data can direct a nurse case manager to the subset of CHF patients likely to benefit from a clinic visit, evaluation, diagnosis, and counseling. This should result in: significantly increased medication compliance, significantly lower emergency department (ED) visits and hospital admissions (both those related to CHF and other conditions related to diminished physical capacity of patients with CHF), and improved physical function.

This study is intended to answer three questions. First, do potentially avoidable acute events (measured by ED visits and hospital admissions) decrease when CHF management is accompanied by systematic telephone-based monitoring as compared with usual care? Second, does medication compliance improve when CHF management is accompanied by systematic telephone-based monitoring as compared with usual care? Third, does perceived health status (physical and emotional function) improve when CHF management is accompanied by systematic telephone-based monitoring as compared with usual care?

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosed CHF
* Member of Kaiser Permanente Georgia

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106
Dates: Start 2001-11; Study Completion 2002-08

PRIMARY OUTCOMES:
Change between study entry and exit (6-months later) in frequency of recommended CHF self-care practices (maintain CHF diary, check weight daily, check ankles and feet for swelling daily)
Knowledge of signs of worsening CHF (sudden weight gain, increase in shortness of breath)
Quality of life

SECONDARY OUTCOMES:
Rate of acute CHF exacerbations (ED visits or hospital admissions for CHF or CHF-related conditions) in the 6-month intervention period compared with the 6-month period preceding study entry.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Roblin, PhD, Principal Investigator — Kaiser Permanente - Georgia Region
Locations (1):
- Kaiser Permanente - Georgia, Atlanta, Georgia, United States